CLINICAL TRIAL: NCT06021340
Title: What To-be-discard Biomaterials From ART Cycles Can Tell us About the Treatment Cycle Outcome?
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Yiu Leung David Chan, Assited Professor, Chinese University of Hong Kong
Other Study IDs: 2023.066
Record Dates: First submitted 2023-08-23; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: IVF; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — IVF cycle to-be-discard biomaterials including follicular fluid, seminal plasma, immature oocytes, abnormal fertilized zygote, unfertilized zygote, arrested embryos, poor quality blastocysts, spent culture medium.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Various to-be-discard material from IVF treatment cycle will be collect and examined, aiming to identify potential reasons of successful outcome or cycle failure.

DETAILED DESCRIPTION:
Usually around 2/3 of IVF material will be discarded at the end of each treatment cycle, including immature oocytes, abnormal fertilized zygotes, poor grading embryos, spent culture medium, etc. Next generation sequencing will be performed for DNA / RNA analysis including the length and the quantity, RNA-seq will be applied for transcriptome profiling, and protein profile will be investigated in a pool sample. By applying various diagnostic tools against those to-be-discard biomaterials, we aim to identify potential underlying reasons of indicating either for an IVF failure or a successful cycle, and try to develop a non-invasive testing method for embryo quality check; better detection of the embryo implantation potential and eventually further increase the IVF clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Assisted Reproductive Technology (ART) Unit of the Chinese University of Hong Kong for ART treatment.
* Participant able to give voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Patient using donor gamete in IVF treatment
* Patient refuses to join and failed to giving consent for any reasons

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population will include patients attending the Assisted Reproductive Technolohy (ART) Unit of the Chinese University of Hong Kong for ART treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
DNA/RNA sequencing data | Through study completion, around 3 year
  DNA / RNA analysis including the length and the quantity, RNA-seq will be applied for transcriptome profiling. Next generation sequencing will be performed to determine the sequence of DNA/RNA for our collected samples.
Proteomic profile | Through study completion, around 3 year
  Protein profile will be investigated in a pool sample, treated samples will go for mass spectrometry (MS) data acquisition and finally destined for data analysis and interpretation.

SECONDARY OUTCOMES:
Blastocyst formation rate | 5 days after fertilization
  Number of blastocysts out of fertilized oocytes observed 5 days after fertilization
Clinical pregnancy rate | Around 5 weeks after embryo transfer
  Clinical pregnancy confirmed by ultrasound
Live birth rate | Around 9 months after embryo transfer
  Birth of a living infant after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Yiu Leung D Chan, DPhil, Principal Investigator — CUHK
Locations (1):
- The Chinese University of Hong Kong and Prince of Wales Hospital, Hong Kong, Hong Kong